CLINICAL TRIAL: NCT01645007
Title: Prevalence of Hepatitis B Infection in the Galilee Region, Israel
Status: Withdrawn | Type: Observational
Why Stopped: The study was not carried out due to lack of funding and budget problems
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0025-12-NHR
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Prevalence; HBsAg; Vaccination; Galilee
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Aims:

1. Evaluate HBV (Hepatitis B Virus) infection prevalence among Druze in the Galilee.
2. Educate the population in order to reduce transmission
3. Increase awareness among primary care providers

Secondary Aims:

1. Identify chronic HBV infected patients who need to be followed and treated,
2. Identify HBV infected women in a childbearing age
3. Identify non immunized individuals and recommend vaccination
4. Identify previously vaccinated individuals who are not immunized
5. Identify previously vaccinated individuals who became infected

Study Design:

Study population is targeted to native Israeli Druze. We aim for evaluating up to 20,000 people from Druze communities in the Galilee area

This work will be divided into three sections:

1. Increasing awareness: lectures and local events will be taken place in the communities. Written information will be given and primary care-providers mainly family doctors, nurses and obstetric surgeons will be involved.
2. All participants, upon signing a consent will:

   * Fill up a questioner
   * Checked for weight, height and waist circumflex
   * Have a blood sample taken
3. Results and recommendations will be forwarded to all participants

ELIGIBILITY:
Inclusion Criteria:

* All consent adults who are 18 year old or older

Exclusion Criteria:

* Individuals younger than 18 year old
* Individuals who cannot or will not sign consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Native Israeli Druze
Sampling Method: Probability Sample
Enrollment: 0 (Actual)